CLINICAL TRIAL: NCT00483054
Title: Efavirenz-based Versus Nevirapine-based Antiretroviral Therapy Among HIV-infected Patients Receiving Rifampin
Acronym: N2R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Collaborators: Mahidol University (Other); Chulalongkorn University (Other)
Responsible Party: Department of Disease Control, Ministry of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210041000824904203
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2009-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; tuberculosis; efavirenz; nevirapine; rifampicin; co-infected HIV and tuberculosis patients
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz (Experimental): Efavirenz 600 mg/day + stavudine +lamivudine
  Interventions: Drug: efavirenz
- Nevirapine (Experimental): Nevirapine 400 mg/day + stavudine +lamivudine
  Interventions: Drug: nevirapine

INTERVENTIONS:
Drug: efavirenz — efavirenz 600 mg/day + stavudine + lamivudine
  Arms: Efavirenz
Drug: nevirapine — nevirapine 400 mg/day + stavudine +lamivudine
  Arms: Nevirapine

SUMMARY:
The randomized controlled trial is conducted among antiretroviral naive co-infected HIV and tuberculosis patients who receiving rifampicin-based antituberculous regimen fro at least 4 weeks butt not exceed 16 weeks before enrolment. All patients receive the same backbone regimen of stavudine (30 mg/40 mg twice daily)+ lamivudie 150 mg twice daily. They are randomized to receive nevirapine 400 mg/day twice daily vs efavirenz 600 mg/day at bed time. All patients are followed through 144 weeks after initiation of antiviral therapy. The primary objective are to compare the proportion of patient who achieve undetectable plasma HIV-1RNA<50 copies/ml at week 48. The previous reports demonstrated that the standard doses of both nevirapine and efavirenz coulde be used among co-infected HIV and tuberculosis patients who receiving rifampicin even though plasma levels are somewhat reduced by rifampicin. However, there have been not been a randomized control trial to compare these two regimens. Thus, this trial will provide the efficacy data between these two regimens.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Positive Serology for HIV-1
* Naïve to antiretroviral therapy
* Baseline CD4 cell counts <250 cells/mm3
* Diagnosed active tuberculosis by clinical features and/or positive acid fast stain and/or positive culture
* Received rifampicin at least 4 weeks but not exceed 16 weeks prior to enrollment
* Willing to participate and sign inform consent

Exclusion Criteria:

* Aspartate transferase enzymes (AST) or alanine transminase enzyme (ALT) >5 times of upper limit
* total bilirubin >3 times of upper limit
* serum creatinine) >2 times of upper limit
* pregnancy or lactation
* receiving immunosuppressive drugs
* receiving any drugs that may have drug-drug interaction with nevirapine and rifampicin
* chronic alcoholic drunken and intravenous drug users
* Previously received single dose of nevirapine to prevent mother to child transmission
* positive for serum cryptococcal antigen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare proportion of patients who achieved undetectable plasma HIV-1RNA< 50 copies/mL at 48 weeks after initiation of antiretroviral treatment between the 2 groups | 48 weeks

SECONDARY OUTCOMES:
to compare CD4 response at 48, 96 and 144 weeks after initiation of antiretroviral treatment, to compare adverse drugs reaction between the 2 groups | 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Manosuthi, MD, Principal Investigator — Bamrasnaradura Infectious Diseases Institute
Locations (1):
- Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi, Thailand

REFERENCES:
- [Derived] Manosuthi W, Sungkanuparph S, Tantanathip P, Lueangniyomkul A, Mankatitham W, Prasithsirskul W, Burapatarawong S, Thongyen S, Likanonsakul S, Thawornwa U, Prommool V, Ruxrungtham K; N2R Study Team. A randomized trial comparing plasma drug concentrations and efficacies between 2 nonnucleoside reverse-transcriptase inhibitor-based regimens in HIV-infected patients receiving rifampicin: the N2R Study. Clin Infect Dis. 2009 Jun 15;48(12):1752-9. doi: 10.1086/599114. PMID 19438397